CLINICAL TRIAL: NCT06383533
Title: An Open-label, Single-arm, Multicenter, Phase II Clinical Study of Disitamab Vedotin Plus Cadonilimab as Therapy in Patients With HER2 Mutant Advanced or Metastatic Bile Duct Adenocarcinoma
Brief Title: Disitamab Vedotin Plus Cadonilimab in Patients With HER2 Mutant Advanced or Metastatic Bile Duct Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-385
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Bile Duct Adenocarcinoma Non-Resectable; HER2 Gene Mutation
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Disitamab Vedotin Plus Cadonilimab (Experimental): Disitamab Vedotin: 2.0mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle. Cardonilimab: 6mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle.
  Interventions: Drug: Disitamab Vedotin Plus Cadonilimab

INTERVENTIONS:
Drug: Disitamab Vedotin Plus Cadonilimab — Disitamab Vedotin: 2.0mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle. Cardonilimab: 6mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle.

SUMMARY:
It is a single arm, open-label, phase II cinical trial to evaluate the efficacy and safety of Disitamab Vedotin Plus Cadonilimab in second-line treatment of patients with Advanced or Metastatic Bile Duct Adenocarcinoma

DETAILED DESCRIPTION:
Biliary tract cancer is a group of highly heterogeneous and aggressive epithelial cancers, accounting for about 3% of all digestive system tumors. It is highly aggressive, and most of them are found in advanced stages, with extremely poor prognosis and a 5-year survival rate of less than 5%. The overexpression rate of HER2 in biliary tract tumors is about 26.5%, and the amplification rate is about 30.1%. In addition, HER2 mutations in biliary tract malignant tumors also include HER2 mutations. In addition, HER2 mutations in biliary malignant tumors also include HER2 mutations. Currently, anti-HER2 strategies have become a new hotspot for exploration in BTC. It is a single arm, open-label, phase II cinical trial conducted in China and plans to recruit 28 patients with HER2 Mutant Advanced or Metastatic Bile Duct Adenocarcinoma who have progressed through first-line treatment. The purpose of this study is to evaluate the efficacy and safety of second-line treatment with Disitamab Vedotin Plus Cadonilimab

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in the study and sign the informed consent;
2. Over 18 years old (including 18 years old), regardless of gender;
3. Expected survival ≥12 weeks;
4. the ECOG physical status score was 0 or 1;
5. For female subjects: they should be surgically sterilized, postmenopausal, or agree to use a medically approved method of contraception (e.g., IUD, birth control pills, or condoms) for the duration of the study treatment and for 6 months after the end of the study treatment period; they must have had a negative blood pregnancy test in the 7 days prior to study drug administration and must not be breastfeeding. For male subjects: should be surgically sterilized or agree to use a medically approved method of contraception during and for 6 months after the end of study treatment;
6. Able to understand the requirements of the trial. Willing and able to comply with the trial and follow-up procedures.
7. Adequate organ function

   1. Bone Marrow Function: (no transfusion within 14 days prior to screening, no use of granulocyte colony stimulating factor [G-CSF], no use of drug correction) : i. Hemoglobin ≥90g/L; ii. Neutrophils ≥1.5×109/L; iii. Platelet ≥100×109/L;
   2. Renal function: calculated creatinine clearance* (CrCl) ≥ 60 mL/min, urine protein < 2+ or 24-hour (h) urine protein quantification < 1.0 g. The Cockcroft-Gault formula will be used to calculate CrCl;

      * The Cockcroft-Gault formula will be used to calculate CrCl CrCL (mL/min) = {(140 - age) × weight (kg) × F}/ (SCr(mg/dL) × 72) where F = 1 for males and F = 0.85 for females; SCr = serum creatinine
   3. liver function: (no albumin infusion within 14 days prior to screening): Serum total bilirubin ≤1.5×ULN (subjects with Gilbert syndrome allow total bilirubin ≤3×ULN) In subjects without liver metastasis, Aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP) ≤2.5×ULN; In subjects with liver metastasis, ALT and AST≤5×ULN, but without elevated bilirubin;
   4. Coagulation function: International Standardized Ratio (INR) and Activated partial thromboplastin time (APTT) ≤1.5 × ULN (unless the subject is receiving anticoagulant therapy and the INR and APTT are within the expected range for treatment with anticoagulants);
   5. Heart function: New York College of Cardiology (NYHA) rating < 3; x. Left ventricular ejection fraction ≥50%;
   6. Nutritional status: (no albumin infusion within 14 days prior to screening): serum albumin ≥ 2.8 g/dL
8. Histologically and/or cytologically confirmed non-treatable locally advanced or metastatic adenocarcinoma of the bile ducts, including intrahepatic or extrahepatic cholangiocarcinoma and gallbladder carcinoma
9. HER2 IHC result of IHC 3+ or IHC 2+, or NGS test suggestive of a HER2 mutation, subject has acceptable prior test results (confirmed by the investigator); or subject is able to provide a specimen from the primary or metastatic site of the tumor wher e the HER2 review/determination was performed;
10. Patients who have progressed or are intolerant to first-line therapy, or whose disease has progressed or recurred during or within 6 months of completion of neoadjuvant/adjuvant therapy
11. The investigator confirmed the presence of at least one measurable lesion according to RECIST 1.1 criteria.
12. Evidence of tumor disease progression or intolerance during or after the most recent treatment as documented by medical history or confirmed by the investigator.

Exclusion Criteria:

Patients who meet any of the following conditions will not be admitted to the study:

1. use of a clinical investigational drug within 4 weeks prior to the start of study treatment;
2. has received major surgical treatment (other than diagnostic) within 4 weeks prior to the start of study treatment and has not fully recovered or is expected to require major surgical treatment during the study;
3. treatment with a live attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of the need for such a vaccine during treatment or within 60 days of the last dose;
4. has had a serious arteriovenous thrombotic event, such as other than cerebrovascular (including transient ischemic attack), deep vein thrombosis, pulmonary embolism, or myocardial infarction, within 6 months prior to study drug administration
5. is suffering from an unstably controlled systemic disease, including diabetes mellitus, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis of the liver, angina pectoris, severe cardiac arrhythmia
6. is suffering from an active infection requiring systemic treatment;
7. a history of active tuberculosis;
8. a positive HIV test result;
9. active HBV or HCV infection; (Note: HBV DNA and/or HCV RNA testing is required for subjects who are HBsAg-positive and/or HCV antibody-positive during the screening period. Subjects who are negative for HBV DNA ≤500 IU/mL (or ≤2000 copies/mL) and/or HCV RNA are eligible for enrollment; HBsAg-positive subjects must be monitored for HBV DNA during the course of treatment).
10. Moderate or severe ascites with clinical symptoms that require therapeutic puncture and drainage (except for small amounts of ascites on imaging without clinical symptoms); uncontrolled or moderate or greater amounts of pleural effusion and pericardial effusion;
11. Known history of severe allergy to any immunosuppressant, anti-HER2 drug;
12. Presence of active autoimmune disease or history of autoimmune disease with potential for relapse (including, but not limited to, autoimmune hepatitis, interstitial pneumonitis, uveitis, enterocolitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism [enrollment is open to subjects who are manageable with hormone replacement therapy only]); subjects with dermatological disorders that do not require systemic therapy such as vitiligo, psoriasis alopecia areata, controlled type I diabetes mellitus treated with insulin or asthma that has completely resolved in childhood and does not require any intervention in adulthood may be enrolled; asthmatics who require medical intervention with bronchodilators may not be enrolled;
13. Patients who, in the judgment of the investigator, have other factors that may affect the results of the study or force the study to be terminated in midstream, such as alcoholism, drug abuse, other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors, which would affect the safety of the patients;
14. Pregnant or breastfeeding women or women/men who are planning to have children;
15. Subjects whose compliance with participation in this clinical trial is estimated to be insufficient or who, in the opinion of the investigator, have other other factors that make them unsuitable for participation in this study;
16. Active malignant tumor other than malignant tumor of the bile duct within 5 years or concurrently. (Except cured limited tumors such as basal cell carcinoma of the skin, squamous carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, and carcinoma in situ of the breast);
17. Tumor lesions with bleeding tendency (e.g., bleeding from ruptured cancerous nodes), history of gastrointestinal bleeding within 6 months prior to the start of study treatment or a definite tendency to gastrointestinal bleeding, e.g., esophagogastric fundal varices at risk for bleeding or severe, locally active peptic ulcer lesions, persistent positive fecal occult blood are not eligible for enrollment (fecal occult blood may be retested if positive at baseline, and if positive at retesting, it requires Gastroduodenoscopy (EGD), or esophagogastric fundal varices if the EGD suggests a risk of bleeding), or blood transfusion 4 weeks prior to study drug administration will be excluded;
18. Patients who are planning to undergo or have previously undergone organ or allogeneic bone marrow transplantation;
19. Subjects with brain metastases and/or carcinomatous meningitis as determined by the Investigator, who have been treated for brain metastases, may be considered for participation in the study if they have been stable for at least 6 months, have not experienced disease progression as determined by imaging within the 4 weeks prior to dosing, and all neurologic symptoms have returned to baseline levels, there is no evidence of new or expanding brain metastases, and they discontinue the use of the drug at least 28 days prior to the first dose of study treatment. No evidence of new or expanding brain metastases and cessation of radiation, surgery, or steroid therapy at least 28 days prior to the first dose of study treatment. This exception does not include carcinomatous meningitis, which should be excluded regardless of whether it is clinically stable;
20. Systemic hormonal therapy for immunosuppression (>10 mg/day of prednisone or other equivalent hormone) within 14 days prior to initiation of study treatment;
21. immunotherapy within 4 weeks prior to the start of study drug administration; chemotherapy (nitrosoureas and mitomycin C within 6 weeks), targeted fractional therapy, or radiotherapy within 2 weeks; and traditional Chinese medicine (traditional Chinese medicine treatments with a clear anti-tumor indication in the specification are eligible for enrollment after a 1-week washout period);
22. Palliative radiotherapy to non-target lesions for symptom control is permitted and must have been completed at least 2 weeks prior to initiation of the study treatment, and radiotherapy-induced adverse events have not recovered to ≤ CTCAE grade 1;
23. Toxicity from prior antineoplastic therapy that has not recovered to CTCAE Grade 0-1, except for: a) alopecia; b) hyperpigmentation; c) peripheral neurotoxicity that has recovered to < CTCAE Grade 2; and d) long-term toxicity due to radiotherapy that, in the judgment of the Investigator, is not recoverable;
24. Liver metastases account for approximately 50% of the entire liver volume;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 12 months
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)

SECONDARY OUTCOMES:
Overall survival (OS) | [Time Frame: up to 36 months]
  The time interval between the start date of study drug and the date of death (any cause)
Progression-free survival (PFS) | [Time Frame: up to 12 months]
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Disease control rate (DCR) | [Time Frame: up to 12 months]
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Incidence of Treatment-Emergent 3/4 Adverse Events | [Time Frame: up to 12 months after enrollment or study close]
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4)

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No